CLINICAL TRIAL: NCT04459676
Title: A Multicenter, Prospective, Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Assess Safety and Efficacy of ANG- 3777 in Patients Hospitalized With Confirmed COVID-19 Pneumonia
Brief Title: Study to Assess Efficacy and Safety Relative to Standard of Care in Patients With COVID-19 Pneumonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Angion Biomedica Corp (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANG3777-ALI-201
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: COVID-19; Pneumonia
Keywords: COVID-19; Acute Lung Injury; Acute Respiratory Distress Syndrome; Pneumonia; Respiratory Failure; AKI
MeSH Terms: conditions — COVID-19; Pneumonia; Acute Lung Injury; Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Standard of Care; terevalefim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ANG-3777 + SOC (Active Comparator): ANG-3777 Administered IV for 30 min and SOC
  Repeat within 24 hours after previous dosing for a total of 4 days
  Interventions: Drug: Standard of Care (SOC) + ANG-3777
- Standard of Care + Placebo (Placebo Comparator): Standard of Care + Placebo
  Interventions: Drug: Standard Of Care (SOC) + Placebo

INTERVENTIONS:
Drug: Standard of Care (SOC) + ANG-3777 — Standard of Care (SOC) + ANG-3777
  Other Names: BB3; Hepatocyte growth factor mimetic
  Arms: ANG-3777 + SOC
Drug: Standard Of Care (SOC) + Placebo — Standard Of Care + Placebo
  Arms: Standard of Care + Placebo

SUMMARY:
To assess the clinical efficacy of ANG-3777 relative to the standard of care in reducing the severity and progression of pulmonary and renal dysfunction and mortality in adult patients hospitalized with COVID-19 pneumonia

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or nonpregnant female 18 years of age or older.
2. Patient has a positive reverse-transcriptase-polymerase-chain-reaction (RT-PCR) assay for SARS-CoV-2 in a respiratory tract sample during the current hospital admission.
3. Patient has pneumonia confirmed by chest imaging.
4. Patient has moderate to severe disease based on the WHO disease severity scale assessment at the time of randomization defined as:

   * Score 4, only those with FiO2 > 40%
   * Score 5 (Non-invasive ventilation or high-flow oxygen)
5. Patient has ability to provide informed consent signed by study patient or legally acceptable representative.
6. Patient has willingness and ability to comply with study-related procedures/assessments

Exclusion Criteria:

1. Has an active malignancy or history of solid or hematological malignancies within 5 years prior to enrollment in the study. Patients who had basal or squamous cell carcinoma-in-situ of the skin that was diagnosed > 2 years prior to the study enrollment and not currently being treated are eligible for study enrollment.
2. Patient is pregnant or breast-feeding.
3. Patient, in the opinion of the investigator, is unlikely to survive for ≥48 hours from the time of screening.
4. Patient has any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study.
5. Patient with alanine aminotransferase (ALT) or aspartate transaminase (AST) > 3x upper limit of normal (ULN) and/or total bilirubin > 2xULN at baseline
6. Patient requires treatment with the cytochrome P450 1A2 (CYP1A2) inhibitors, ciprofloxacin (Cipro®) and/or fluvoxamine (Luvox®)
7. Patients participating in any other clinical trial with an investigational drug product or procedure
8. Recipients of solid organ and/or hematopoietic cell transplantation
9. Patient is known to have End Stage Renal Disease (ESRD) and was being treated with maintenance hemodialysis or peritoneal dialysis prior to the current hospitalization.

Note: Patients who initiated RRT due to Acute Kidney Injury during their current hospitalization will be eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients alive, without the need for mechanical ventilation and free of the need for RRT (on an ongoing basis) at Day 28 | From the time of randomization until (Day 1) until death or until Day28, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: John Neylan, MD, Study Director — Angion Biomedica
Locations (10):
- Brazil (10):
  - Hospital Vera Cruz - NUPEC Nucleo de Pesquisa Clínica, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Pontifícia Universidade Catolica de Campinas, Campinas, São Paulo
  - UPCLIN - Faculdade de Medicina da UNESP Campus de Botucatu, Botucatu
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (HCFMRP), Ribeirão Preto
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital Heliópolis-SP, São Paulo
  - Hospital Vila Nova Star, São Paulo
  - Irmandade da Santa Casa de Misericórdia de São, São Paulo
  - Santa Casa de Misericordia de Sao Paulo, São Paulo